CLINICAL TRIAL: NCT00082446
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of MVA-BN in a Dose Response Regimen Followed by Administration of Dryvax in Healthy Adult Volunteers
Brief Title: Combination Study With MVA BN and Dryvax
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 02-017; POX-MVA-002
Record Dates: First submitted 2004-05-10; First posted 2004-05-11 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2008-09

CONDITIONS: Smallpox
Keywords: Smallpox, vaccine
MeSH Terms: conditions — Smallpox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- E (Experimental): Subject will receive an SC dose of MVA 1x10^8 on day 0 and day 28. On day 112 subjects will receive a dose of placebo by scarification.
  Interventions: Biological: MVA Smallpox Vaccine; Other: Placebo
- D (Active Comparator): Subject will receive a SC dose of placebo on day 0 and day 28. On day 112 subjects will receive a dose of Dryvax® by scarification.
  Interventions: Biological: Live vaccinia virus vaccine; Other: Placebo
- C (Experimental): Subject will receive a SC dose of MVA 1x10^8 on day 0 and day 28. On day 112 subjects will receive a dose of Dryvax® by scarification.
  Interventions: Biological: Live vaccinia virus vaccine; Biological: MVA Smallpox Vaccine
- B (Experimental): Subjects will receive a SC dose of MVA 5x10^7 on day 0 and day 28. On day 112 subjects will receive a dose of Dryvax® by scarification.
  Interventions: Biological: Live vaccinia virus vaccine; Biological: MVA Smallpox Vaccine
- A (Experimental): Subjects will receive a SC dose of MVA 2x10^7 on day 0 and day 28. On day 112 subjects will receive a dose of Dryvax® by scarification.
  Interventions: Biological: Live vaccinia virus vaccine; Biological: MVA Smallpox Vaccine
- F (Experimental): Subject will receive an IM dose of MVA 1x10^8 on day 0 and day 28. On day 112 subjects will receive a dose of Dryvax® by scarification.
  Interventions: Biological: Live vaccinia virus vaccine; Biological: MVA Smallpox Vaccine

INTERVENTIONS:
Biological: Live vaccinia virus vaccine — Dryvax®: 0.25 mL of vaccine will be administered by the standard route of scarification using a bifurcated needle on day 112 for Groups A, B, C, D and F.
  Arms: A; B; C; D; F
Biological: MVA Smallpox Vaccine — Imvamune/MVA-BN 1x10^8 will be administered intramuscularly to Group F on day 0 and day 28.
  Arms: F
Biological: MVA Smallpox Vaccine — Imvamune/MVA-BN Groups A, B C and E will be administered subcutaneously: 2x10^7, 5x10^7, 1x10^8, 1x10^8, respectively, on days 0 and day 28.
  Arms: A; B; C; E
Other: Placebo — Group E will receive sterile saline placebo for injection via scarification on day 112.
  Arms: E
Other: Placebo — Group D will receive sterile saline placebo for injection subcutaneously on day 0 and day 28.
  Arms: D

SUMMARY:
The overall goals of this study are to expand the available data on the safety and immunogenicity of MVA-BN in vaccinia-naive adults and to determine the optimum dose of MVA-BN to induce immune responses and attenuate Dryvax take reactions. Participants will include 90 healthy volunteers, ages 18-32 years. Participants will be randomly assigned to 1 of 6 study groups (groups A-F). Participants will be involved in study related procedures for up to 2 years. During this time, volunteers will return periodically for blood draws to check immune responses.

DETAILED DESCRIPTION:
The primary goal of this phase I trial is to expand the available data on the safety and immunogenicity of MVA-BN in vaccinia-naïve adults. The secondary goals of this vaccine trial are: to determine the optimum dose of MVA-BN, given twice, to induce an immune response and attenuate Dryvax® take reactions; and to compare the ability of 2 routes of administration of MVA-BN, subcutaneous and intramuscular, to induce an immune response at the highest tested dose. A total of 90 healthy adult volunteers ages 18-32 will participate in this study. The volunteers will be randomly assigned to 1 of 6 groups to be immunized with: MVA-BN (subcutaneously) at 1 of 3 dose levels and Dryvax® (per scarification); placebo (subcutaneously) and Dryvax® (per scarification); MVA-BN (subcutaneously) at the highest dose level and placebo scarification; or MVA-BN (intramuscularly) at the highest dose level and Dryvax® (per scarification). The study will last about 30 months. Each volunteer's participation will last 6 months for all treatment groups. Subjects randomized to treatment groups D and E will have follow-up for 2 years. During this time, volunteers will return periodically for blood draws to check immune responses. Subjects will require visits for dressing changes as needed post-Dryvax vaccination. Variables to be investigated include: adverse events and side effects to the vaccines, and immunogenicity testing including antibody and cellular responses to the vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-32.
* Never received smallpox vaccination.
* Read, signed and dated informed consent document.
* Availability for follow-up for the planned duration of the study two years after first immunization.
* Acceptable medical history by screening evaluation and limited physical examination.
* For women, negative serum pregnancy test at screening and negative urine or serum pregnancy test within 24 hours prior to vaccination.
* If the volunteer is female and of child bearing potential, she agrees to use acceptable contraception, and not become pregnant for at least 56 days after the last vaccination. A woman is considered of child bearing potential unless post-menopausal or surgically sterilized. [Acceptable contraception methods are restricted to effective intrauterine devices (IUDs) or licensed hormonal products with use of method for a minimum of 30 days prior to vaccination.] Women who are not sexually active must agree to use one of the acceptable contraception methods if they are of childbearing potential.
* Negative ELISA for HIV.
* ALT<1.25 times institutional upper limit of normal.
* Negative hepatitis B surface antigen and negative antibody to hepatitis C virus.
* Negative urine glucose by dipstick or urinalysis.
* Adequate renal function defined as a serum creatinine less than or equal to 1.4mg/dL for males and less than or equal to 1.2mg/dL for females; urine protein < 30 mg/dL or none or trace proteinuria (by urinalysis or dipstick); and a calculated creatine clearance greater than or equal to 80 mL/min. based on the following formulas:
* Males [(140-age in years) X weight in kg]/(72 X serum creatinine)
* Females 0.85X[(140-age in years) X weight in kg]/(72 X serum creatinine)
* ECG without clinical significance (e.g., all kinds of atrioventricular or intraventricular conditions or blocks such as complete left or right bundle branch block, AV-node block, QTc or PR prolongation, premature atrial contractions or other atrial arrhythmia, sustained ventricular arrhythmia, or 2 premature ventricular contractions (PVC) in a row, or ST elevation consistent with ischemia)
* CBC: Hemoglobin >11g/dl; White blood cells greater than 2,500 and less than 11,000/cubic mm; Platelets greater than or equal to 140,000/cubic mm.

Exclusion Criteria:

* History of immunodeficiency.
* Typical vaccinia scar.
* Known or suspected history of smallpox vaccination.
* Military service prior to 1989 or after January 2003.
* Known or suspected impairment of immunologic function including, but not limited to, clinically significant liver disease; diabetes mellitus; moderate to severe kidney impairment.
* Malignancy, including squamous cell skin cancer or basal cell skin cancer at vaccination site or history of skin cancer at the vaccination site.
* Active autoimmune disease. Persons with vitiligo or thyroid disease on thyroid replacement are not excluded.
* History of keloid formation.
* History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, or other heart condition under the care of a doctor.
* History of an immediate family member (father, mother, brother or sister) who has had onset of ischemic heart disease before age 50 years.
* Ten percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's Risk Assessment Tool for Estimating Your 10-Year Risk of Having a Heart Attack, located at the following URL: http://hin.nhlbi.nih.gov/atpiii/calculator.asp. NOTE: This criterion applies only to volunteers 20 years of age and older.
* Abnormal troponin I.
* Use of immunosuppressive medication. Corticosteroid nasal sprays are permissible. Persons who have used topical steroid can be enrolled after their therapy is completed.
* Medical or psychiatric condition or occupational responsibilities that preclude volunteer compliance with the protocol.
* Any history of "illegal" injection drug use.
* Receipt of inactivated vaccine 14 days prior to vaccination.
* Receipt of live attenuated vaccines within 30 days of vaccination.
* Use of experimental agents within 30 days prior to vaccination.
* Receipt of blood products or immunoglobulin in the 6 months prior to vaccination.
* Acute febrile illness (greater than or equal to 100.5 degrees F) on the day of vaccination.
* Pregnant or lactating women.
* Eczema of any degree or history of eczema.
* People with atopic dermatitis, Varicella zoster, chronic exfoliative skin disorders/conditions or any acute skin disorders of large magnitude, e.g., laceration requiring sutures, burn greater than 2x2 cm.
* Household contacts/sexual contacts with, or occupational exposure to (other than minimal contact), any of the following: Pregnant women; Children <12 months of age; People with or history of eczema; People with atopic dermatitis, Varicella zoster, chronic exfoliative skin disorders/conditions or any acute skin disorders of large magnitude, e.g., laceration requiring sutures, burn greater than 2x2 cm; People with immunodeficiency disease or use of immunosuppressive medications.
* Any condition that, in the opinion of the investigator, might interfere with study objectives.
* Known allergies to or any component of MVA or MVA-BN vaccine (e.g., tris(hydroxymethl)-amino methane, sodium chloride, sucrose, dextran, L-Glutamic acid monopotassium, chicken embryo fibroblast proteins, gentamycin).
* Known allergy to egg or aminoglycoside.
* Known allergies to any component of the Dryvax® vaccine (e.g. polymyxin B sulfate, dihydrostreptomycin sulfate, chlorotetracycline hydrochloride, neomycin sulfate).
* Known allergies to any known component of the Dryvax® diluent (i.e. glycerin and phenol).
* Known allergies to any known components of vaccinia immunoglobulin (VIG), i.e. thimerosal or previous allergic reaction to immunoglobulins.
* Known allergies to cidofovir or probenecid.
* Study personnel.

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2004-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Adverse Events and side effects to the vaccines. | Reactogenicity will be evaluated for a 2-week period post-vaccination at each time point and for the duration of study.

SECONDARY OUTCOMES:
Immunogenicity testing of antibody and cellular responses to the vaccines. | Visit days 0, 14, 28, 42, 56, 112, 140, 182, 365, and 730.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

REFERENCES:
- [Result] Elizaga ML, Vasan S, Marovich MA, Sato AH, Lawrence DN, Chaitman BR, Frey SE, Keefer MC; MVA Cardiac Safety Working Group. Prospective surveillance for cardiac adverse events in healthy adults receiving modified vaccinia Ankara vaccines: a systematic review. PLoS One. 2013;8(1):e54407. doi: 10.1371/journal.pone.0054407. Epub 2013 Jan 17. PMID 23349878